CLINICAL TRIAL: NCT04749485
Title: A Single-armed Open-labeled Phase II Study of HX008 (a Humanized Monoclonal Antibody Targeting PD-1) for the Treatment of Patients With Locally Advanced or Metastatic Melanoma Who Have Failed the Standard Treatments.
Brief Title: A Study of HX008 for the Treatment of Patients With Malignant Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX008-II-MM-01
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HX008 (Experimental)
  Interventions: Drug: HX008

INTERVENTIONS:
Drug: HX008 — Patients will receive HX008 3mg/kg by intravenous (IV) infusion on Day 1, every 3 weeks (Q3W), till progressed disease or withdrawal.

SUMMARY:
HX008 is a humanized monoclonal antibody targeting PD-1 on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors. In this study, the efficacy and safety of HX008 in patients with locally advanced or metastatic melanoma who have failed the standard treatments will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent voluntarily. Understand this protocol and be willing and able to adhere to the study visit schedule;
* Male and Female aged 18 to 75 are eligible;
* Histologic diagnosis of locally advanced unable to undergo complete resection or metastatic melanoma, while ocular melanoma is excluded, and the overall rate of mucosal melanoma is no more than 22%.
* Has failed at least 1 prior routine regimen for advanced disease, including chemotherapy, target therapy, immunotherapy, biological therapy (IFN-gamma, interleukin, onco-vaccine, cytokine, oncolytic virus or cancer growth factor inhibition), and the interval between last previous treatment and the first dose of this trial should be ≥ 4 weeks or 5 half-life of the previously administrated drug, which happens first.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Life expectancy ≥ 3 months.
* At least 1 measurable extracranial lesion based on RECIST v1.1, and no prior radiation to measurable lesions;
* Central nervous system metastases must be asymptomatic with or without treatment, and be stable for at least 3 months based on CT/MRI, and no need for systemic steroids within 4 weeks prior to the first dose of the study drug.
* Providing with tumor specimen (for testing the expression of PD -L1);
* Has sufficient organ and bone marrow function to meet the following laboratory examination standards: neutrophils ≥ 1.5 x 10^9/L; white blood cells ≥3.0 x 10^9/L; platelets ≥ 100 x 10^9/L; hemoglobin ≥ 90 g/L; serum creatinine ≤1x ULN; aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; total bilirubin ≤ 1.5 x ULN; INR≤2 x ULN, aPTT≤1.5 x ULN (except for those undergoing anticoagulant therapy);
* Reproductive men and women of childbearing age are willing to take effective contraceptive measures from signing the informed consent form to 3 months after the last administration of the trial drug.

Exclusion Criteria:

* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as carcinoma in situ of the cervix or basal cell skin cancer.
* With adverse reactions of previous treatment that have not recovered to CTCAE V5.0 grade ≤ 1, except for the residual hair loss effect.
* Prior treatment with anti-PD-1/PD-L1/CTLA-4 antibody.
* With active or history of autoimmune diseases that may recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulitis, etc.), or patients with high risk (e.g., organ transplantation requiring immunosuppressive therapy). While those with the following diseases were allowed to be enrolled: a) Stable patients with type I diabetes after a fixed dose of insulin; b) Autoimmune hypothyroidism requiring hormone replacement therapy only; c) Skin diseases requiring no systemic treatment (e.g. eczema, skin rash covering less than 10% of the body surface, psoriasis without ophthalmic symptoms, etc.).
* Expecting to receive major surgery during the study period including 4 weeks prior to the first dose of the study drug.
* Need to receive systemic corticosteroids (dose equivalent to > 10 mg prednisone / day) or other immunosuppressive drugs within 14 days before enrollment or during the study period. Those under the following conditions are eligible: a) Locally external use or inhaled corticosteroids; b) short-term (≤ 7 days) use of glucocorticoids for the prevention or treatment of non-autoimmune allergic diseases.
* History of human immunodeficiency virus infection, acquired or congenital immunodeficiency disease, organ transplantation or stem cell transplantation.
* Has active chronic HBV or HCV infection, except those with HBV DNA viral load ≤500 IU/mL or <10^3 copies/mL, or HCV RNA negative after adequate treatment.
* Has severe infection within 4 weeks or active infection requiring IV infusion or oral administration of antibiotics within 2 weeks prior to the first dose of the study drug.
* Known to be allergic to macromolecular protein agents or monoclonal antibody; Known to has a history of severe allergies to any of the components in the study drug (CTCAE v5.0 ≥ grade 3);
* Has participated in other clinical trial within 4 weeks prior to the first dose of the study drug.
* Alcohol dependence or drug abuse within recent one year.
* Has a history of confirmed neurological or mental disorders, such as epilepsy, dementia; or with poor compliance; or the presence of peripheral neurological disorders.
* Has brain metastasis with symptoms.
* Is pregnant or breastfeeding.
* Other reasons disqualifying the entering of this study based on the evaluation of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2021-11-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 36 months

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  Progression-free survival (PFS) is defined as the time from the first study drug treatment to disease progression (PD) or to death of the subject due to any reason.
Duration of Response (DOR) | 24 months
  Duration of Response (DOR) is defined as the time from the first evidence of response (PR or CR) to the first evidence of PD or the date of death for any reason.
Overall survival (OS) | 36 months
  Overall survival (OS) refers to the time from the first study drug treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Study Chair — Peking University Cancer Hospital and Research Institute
Locations (11):
- China (11):
  - Peking University Cancer Hospital and Research Institute, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The first Hospital of Jilin University, Changchun, Jilin
  - Fudan Universtiy Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan Universtiy, Chengdu, Sichuan
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang University School of Medicine Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Cui C, Chen Y, Luo Z, Zou Z, Jiang Y, Pan H, Fan Q, Zhao J, Xu Q, Jiang R, Wang X, Ma T, Guo Z, Si L, Chi Z, Sheng X, Dou Y, Tan Q, Wu D, Guo J. Safety and efficacy of Pucotenlimab (HX008) - a humanized immunoglobulin G4 monoclonal antibody in patients with locally advanced or metastatic melanoma: a single-arm, multicenter, phase II study. BMC Cancer. 2023 Feb 6;23(1):121. doi: 10.1186/s12885-022-10473-y. PMID 36747118